CLINICAL TRIAL: NCT04200066
Title: A Phase 1 Study of Maprotiline in Combination With Tamoxifen and Temozolomide for Recurrent Glioblastoma
Brief Title: A Study of Maprotiline in Combination With Tamoxifen and Temozolomide for Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: One of the drugs for the study is not commercially available.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nimish Mohile, Associate Professor of Neurology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBRT19062
Record Dates: First submitted 2019-12-05; First posted 2019-12-16 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Glioblastoma; Brain Tumor
Keywords: Maprotiline; Tamoxifen; Temozolomide
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Temozolomide; Tamoxifen; Maprotiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): This arm will combine maprotiline with temozolomide and tamoxifen to determine the maximum tolerated dose.
  Interventions: Drug: Temozolomide, Tamoxifen, Maprotiline

INTERVENTIONS:
Drug: Temozolomide, Tamoxifen, Maprotiline — Subjects will receive a combination of temozolomide and tamoxifen for two weeks. After that, they will receive a combination of temozolomide, tamoxifen and maprotiline for the remainder of the study. All drugs are administered orally. Subjects will undergo visits at the beginning of week 3, week 5 and week 7 that will involve multiple blood draws and ECGs to evaluate for pharmacokinetics and drug interactions. Response will be assessed every two months with an MRI and patients will continue on study as long as their tumors are under control and they are tolerating the regimen.
  Other Names: TMZ; TMX; TMT

SUMMARY:
The main purpose of this study is to find out the highest possible dose of maprotiline that can be given safely in combination with temozolomide and tamoxifen.

DETAILED DESCRIPTION:
The main purpose of this study is to find out the highest possible dose of maprotiline that can be given safely in combination with temozolomide and tamoxifen. Temozolomide is approved to treat glioblastoma and the investigator wants to understand what doses are safe to use. Tamoxifen has been used for many years to treat breast cancer and there have also been studies combining it with temozolomide for the treatment of brain tumors that have shown the combination to be safe. In this study, the investigator will be adding maprotiline to temozolomide and tamoxifen, determining the highest possible dose that is safe, making sure there are no significant drug interactions and studying the safety of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven World Health Organization (WHO) grade IV gliomas. Patients will be eligible if the original histology was a grade II or grade III glioma as long as a subsequent histological diagnosis of a grade IV glioma is confirmed.
* Patients must have undergone upfront therapy that included a combination of radiotherapy and concurrent and adjuvant temozolomide.
* Patients must have shown unequivocal radiographic evidence for tumor progression by MRI scan. A scan should be performed within 10 days prior to registration and on a steroid dose that has been stable for at least five days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI is required.
* Patients must have tissue confirmation of histology at the University of Rochester
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery (including gamma-knife or cyber-knife) must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy, MR Perfusion, or surgical documentation of disease. The decision of which modality to use to make this confirmation will be at the discretion of the investigator.
* Patients who have undergone re-resection for recurrent disease are eligible but must have an interval of 7 days prior to starting therapy.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
* Age > 18 years old, and with a life expectancy > eight weeks.
* Karnofsky Performance Status ≥ 70
* Patients must have an interval of at least 28 days from any investigational agent or from prior cytotoxic therapy, six weeks from prior nitrosureas, three weeks from procarbazine and two weeks from vincristine.
* Patients must have failed prior radiotherapy and must have an interval of greater than 90 days from completion of initial radiation therapy to study entry.
* WBC > 3,000/µl, ANC > 1,500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 8 gm/dl). Patients must have adequate liver function (SGOT and bilirubin < 1.5 times ULN), and adequate renal function (creatinine clearance >30ml/min as measured by Cockroft-Gault formula) <before starting therapy. These tests must be performed within 2 weeks prior to treatment initiation. Eligibility level for hemoglobin may be reached by transfusion.
* Patients with any number of recurrences are eligible.
* Patients taking tamoxifen for other indications are eligible for the study

Exclusion Criteria:

* Patients who are within 3 months of treatment with radiation and concurrent temozolomide will not be eligible unless there are new enhancing abnormalities outside the high dose radiation fields (i.e. beyond the 80% isodose line) or surgical demonstration of active tumor.
* Patients must not be pregnant and must agree to practice adequate contraception. Women of childbearing potential must have a negative B-HCG pregnancy test documented within 7 days prior to registration. Women must not be breastfeeding.
* Patients with a history of other cancer (except non-melanoma skin cancer or cancer of the cervix), unless in complete remission for at least three years are ineligible.
* Concomitant use of enzyme inducing anti-epileptic drugs will be prohibited. These include phenytoin, phenobarbital, carbamazepine and oxacarbazepine. If patients are on these at time of study enrollment, drugs can be transitioned to a non-enzyme inducing anti-epileptic drug at the discretion of the investigator.
* Patients must not have any significant medical illnesses or other history that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have concurrent use of other tricyclic antidepressants or MAO inhibitors.
* Patients with lower urinary tract symptoms secondary to benign prostatic hypertrophy that are refractory to medications
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
* Patients with history of myocardial infarction within the past year.
* Patients with prior history of status epilepticus
* Patients with evidence of QTc prolongation greater than 450ms
* Patients receiving strong CYP2D6 inhibitors (bupropion, fluoxetine, paroxetine, quinidine, terbinafine) will be excluded.
* Patients receiving strong CYP3A4 inhibitors (Clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir) will be excluded.
* Patients with history of hypersensitivity to maprotiline.
* Patient meets the cut-off score of ≥ 12 in the PHQ-9 or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dosing Regimen (MTDR) of maprotiline in combination with temozolomide (TMZ) and tamoxifen (TMX) | through study completion, an average of 6 months
  Assessment of toxicity based on the NCI common toxicity criteria.

SECONDARY OUTCOMES:
Mean Maprotiline drug level | week 7
  Blood sampling for pharmacokinetic assessment of study drugs. The mean maprotiline drug level will be reported. The drug levels will be measured at 2, 5, and 7 hours on weeks 1, 2, 3, 5 and 7
Median Maprotiline drug level | week 7
  Blood sampling for pharmacokinetic assessment of study drugs. The median maprotiline drug level will be reported. The drug levels will be measured at 2, 5, and 7 hours on weeks 1, 2, 3, 5 and 7
6 mo Progression Free Survival | 6 months
  Measure of time from study enrollment until progression.
  Progressive Disease: >25% increase in the bi-dimensional area OR an increase in T2/FLAIR abnormality that is consistent with tumor OR the presence of a new lesion OR clinical deterioration.
Overall Survival | from date of enrollment until date of death from any cause up to 60 months
  Measure of time from study enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nimish Mohile, MD, Principal Investigator — University of Rochester